SEMALCO study Statistical Analysis Plan EU CT NUMBER: 2023-503371-25-00

Edition: 1.0

03.06.25

# SEMALCO- Statistical Analysis Plan

Does the Glucagon-like Peptide 1 (GLP-1) receptor agonist semaglutide reduce alcohol intake in patients with alcohol use disorder and comorbid obesity?

EU CT NUMBER: 2023-503371-25-00 Clinicaltrials.gov: NCT05895643 UTN-NUMBER: U1111-1286-6919

SAP date/status 03.06.25/ 1<sup>st</sup> edition

Protocol version: 28.06.23/ 3<sup>rd</sup> edition

SAP CONTRIBUTORS:

#### SPONSOR-INVESTIGATOR

Anders Fink-Jensen MD DMSc Professor Psychiatric Centre Copenhagen, Frederiksberg University of Copenhagen, Denmark

### **INVESTIGATOR**

Mette Kruse Klausen MD, PhD
Postdoc
Psychiatric Centre Copenhagen, Frederiksberg

#### **SENIOR STATISTICIAN RESPONSIBLE**

Claus Thorn Ekstrøm PhD
Professor
Section of Biostatistics
University of Copenhagen, Denmark

#### STATISTICIAN RESPONSIBLE

Andreas Jensen PhD
Senior researcher
Department of Paediatrics and Adolescent Medicine, Rigshospitalet

SEMALCO study Statistical Analysis Plan EU CT NUMBER: 2023-503371-25-00

## Psychiatric Centre Copenhagen, Frederiksberg Hospital

03.06.25 Edition: 1.0

| Signatures: | |
|---------------------|---------|
| Anders Fink-Jensen | |
| | _ Date: |
| Claus Thorn Ekstrøm | |
| | Date: |
| Mette Kruse Klausen | |
| | _ Date: |
| Andreas Jensen | |
| | Date: |

03.06.25

Edition: 1.0

EU CT NUMBER: 2023-503371-25-00

Abbreviations

Statistical Analysis Plan

**SEMALCO** study

AUD

AUDIT Alcohol use disorder identification test

BOLD-response Blood-oxygen-level-dependent response

CBT Cognitive behavioral therapy

DSM-5 Diagnostic and Statistical Manual of Mental Disorders

Alcohol Use Disorder

DTI Diffusion tension imaging

fMRI Functional magnetic resonance imaging (brain-scan)

GABA gamma-aminobutyric acid

GLP-1RA Glucagon-like peptide-1 receptor agonist

Heavy drinking day Alcohol consumption over 60/48 g (men/women) of alcohol per day

ICD-10 International Classification of Diseases

MRS Magnetic Resonance Spectroscopy

PEth Phosphatidylethanol - Biomarker for alcohol consumption

RCT Randomised clinical trial

REDCap Web application for building and managing online surveys and databases

TLFB Time-Line-Follow-Back Method (recording of heavy drinking days)

WHO World Health Organization

EU CT NUMBER: 2023-503371-25-00

# Table of content

| Abbreviations | 3 |
|---|---|
| Introduction | <u>5</u> 6 |
| Hypotheses | <u>6</u> 7 |
| Study Methods | <u>6</u> 7 |
| Trial design | <u>6</u> 7 |
| Randomisation | <u>6</u> 7 |
| Sample size | <u>7</u> 8 |
| Framework, Statistical interim analysis and stopping guidance | <u>7</u> 8 |
| No superiority, equivalence, or noninferiority hypothesis testing framework was performed. | <u>7</u> 8 |
| Timing of final analysis | <u>7</u> 8 |
| Timing of outcome assessments | <u>7</u> 8 |
| Statistical Principles | <u>8</u> 9 |
| Confidence intervals and P-values | <u>8</u> 9 |
| Adherence and protocol deviations | <u>8</u> 9 |
| Analysis populations | <u>8</u> 9 |
| Trial Population | <u>8</u> 9 |
| Screening data | <u>8</u> 9 |
| Eligibility | <u>8</u> 9 |
| Recruitment | <u>9</u> 10 |
| Withdrawal/Follow up | <u>9</u> 10 |
| Baseline Patient characteristics | <u>9</u> 10 |
| Analysis | <u>10</u> 11 |
| Primary endpoint | <u>10</u> 11 |
| Secondary endpoints | <u>10</u> 11 |
| Descriptive statistics | <u>11</u> <del>12</del> |
| Analysis methods | <u>11</u> <del>12</del> |
| Missing data/sensitivity analysis | <u>12</u> 13 |
| Subgroup analysis | <u>12<del>13</del></u> |
| Tertiary analyses | <u>12</u> 13 |
| Harms | <u>13</u> 14 |
| Statistical software | <u>13</u> 14 |
| References | <u>14<del>15</del></u> |

**SEMALCO** study Statistical Analysis Plan

EU CT NUMBER: 2023-503371-25-00

03.06.25 Edition: 1.0

## Introduction

Alcohol use disorder (AUD) is a chronic brain disorder characterised by loss of control of alcohol intake, a negative state when not consuming alcohol, and compulsive alcohol behaviour, leading to relapse. Globally, alcohol use is a huge burden, and an estimated 280 million people globally suffer from AUD.<sup>2</sup> In 2016, three million deaths were caused by the harmful use of alcohol. In Denmark, 14% of the Danish population has a harmful consumption of alcohol, and 3% fulfils the criteria for AUD.<sup>3</sup> Despite this, the treatment gap is wide compared to other mental health disorders<sup>4</sup> - a Danish study has reported an all-cause cumulative 15-year mortality rate of 29% after a first-time hospital contact due to alcohol.<sup>5</sup> This high mortality rate might be due to medical conditions and complications such as alcoholic liver disease, injuries, <sup>1</sup> fracture, <sup>5</sup> heart disease, stroke, cancer,<sup>6</sup> or suicide.<sup>7</sup> In this perspective, AUD has serious consequences for the individual, families and friends<sup>6</sup> and the society due to higher health care<sup>5</sup> and socio-economical costs.<sup>2,8</sup> This is also why alcohol is reported as the most harmful drug of addiction; the harm to both users and others taken into consideration.<sup>9</sup>

One of the best-documented modalities in the treatment of AUD is cognitive-behavioural therapy (CBT). 10-12 The underlying neuroanatomical basis of alcohol addiction and treatment effects of CBT are not yet established, though functional Magnetic Resonance Imaging (fMRI) studies have begun to elucidate the neuroanatomical basis. The pharmacological treatment of AUD is considered an important supplement to psychological therapy. Disulfiram, 13 a substance that blocks alcohol-metabolising enzymes resulting in increased acetaldehyde concentrations, was introduced in Denmark many years ago and is still the most used drug against AUD in Denmark. Newer pharmacological agents such as acamprosate<sup>13</sup> and naltrexone<sup>13</sup> have been introduced to the clinic. However, despite numerous randomised clinical trials (RCT), these compounds have not gained widespread dissemination, probably because the effect of these substances has been modest, with a less than 10% increase in abstinent rate compared to placebo.

As the success rates of CBT are moderate and the synergistic effects of adding pharmacological treatment – as described above – are quite limited, strong needs still exist for efficient, molecular targets in the medical treatment of alcohol use disorder.14

GLP-1-based therapy was introduced to the market in 2006, and since then, several GLP-1 (GLP-1RAs) have been approved for treating type 2 diabetes and/or obesity. The proposed GLP-1RA semaglutide is reported to be superior to previous GLP-1 RAs approved for weight loss, 15 and was approved by the FDA to treat obesity in June 2021 (Wegovy®). Several pre-clinical studies report of GLP-1RAs crossing the blood-brain

03.06.25

Edition: 1.0

SEMALCO study Statistical Analysis Plan

EU CT NUMBER: 2023-503371-25-00

barrier to some extent, 16-19 and semaglutide is reported to access the brainstem, septal nucleus, and

hypothalamus.16

Several GLP-1RAs have been evaluated in pre-clinical addiction models regarding their effects on alcohol

consumption in mice, rats, and nonhuman primates. Also, register-based cohort studies, brain imaging, and

preliminary clinical data indicate that GLP-1RAs could be a potential new treatment for AUD.<sup>20</sup> However,

larger RCTs are needed to investigate whether these beneficial findings on alcohol consumption can be

extended to encompass patients with known alcohol use disorder.<sup>21</sup>

Hypotheses

Treatment with semaglutide will:

• Cause a greater decrease in alcohol consumption compared with placebo, measured as the total

number of heavy drinking days, in patients with AUD and comorbid obesity

Cause a reduced fMRI BOLD response compared with placebo in reward processing regions (ventral

and dorsal striatum, putamen, nucleus accumbens, and caudate), including the septal area

• Cause a greater increase in brain GABA levels compared with placebo, measured with an MRS scan

Study Methods

Trial design

The SEMALCO trial is a 26-week, randomised, double-blinded, placebo-controlled clinical trial.<sup>22</sup> Comparative

treatment regimens were once-weekly injections with semaglutide 2.4 mg (Wegovy®) or placebo (saline) as

a supplement to cognitive behavioural therapy. Baseline data were collected at the screening session. Follow-

up meetings were scheduled at weeks 6, 8, 12, 16, 20, and a final evaluation at week 26. A subgroup of

patients had a combined baseline fMRI- and MRS scan performed before receiving their first injection and

again when finalising the study.

Randomisation

The participants were randomised into two groups: semaglutide or placebo. The randomisation was stratified

in terms of age, sex, and baseline alcohol consumption, i.e., the number of heavy drinking days in the

recorded 30 days before inclusion measured by the TLFB method (6-11, 12-17, 18-23, 24-30 days). The

randomisation tool in REDCap was used for this stratified randomisation. Patients, investigators, other

03.06.25

Edition: 1.0

SEMALCO study Statistical Analysis Plan

EU CT NUMBER: 2023-503371-25-00

caregivers performing assessments, and persons performing data analysis were blinded from the time of

randomisation until the time of database unlock. To maintain the blinding, the participants were blindfolded,

and as the active pen made a small sound when released, the patients were also provided with music in their

ears. An un-blinded nurse prepared the injection in a separate room and gave the injection immediately after.

Sample size

The sample size calculation was based on the primary endpoint, i.e., the change in heavy drinking days from

baseline to end of follow-up (week 26). No other studies have investigated the effects of semaglutide in

treatment-seeking patients with alcohol use disorder. The sample size calculation is thus based on the alcohol

study by Bogenschutz et al., 23 investigating psilocybin-assisted psychotherapy as a novel treatment of AUD.

They reported a reduction in the total number of heavy drinking days of 46.77% in the intervention group

and 25% in the placebo group. With a power of 90%, an alpha of 5%, and an estimated standard deviation

(SD) of 26.44, a total of 64 patients, 32 patients in each treatment group, is needed. Large drop-out rates are

often observed in AUD intervention trials, with attrition rates between 10% and 35%.<sup>24</sup> Assuming a 40% drop-

out rate, the total required sample size is 108, with 54 patients in each treatment group. All patients will be

included at one research site (Psychiatric Centre Copenhagen, Frederiksberg Hospital).

Framework, Statistical interim analysis and stopping guidance

No superiority, equivalence, or noninferiority hypothesis testing framework was performed.

No interim analysis was performed.

Timing of final analysis

All analyses will be carried out with the treatment groups still blinded and labelled as "Treatment Group A1"

and "Treatment Group B2". Before dividing participants into "group A-1" and "group B2", the statistical

analysis plan will be completed, signed, and uploaded at ClinicalTrials.gov, and the data set locked. The final

unblinding of treatment groups (semaglutide or placebo), will not be carried out until all statistical analyses

are performed.

Post-hoc analyses, if performed, will be conducted unblinded.

Timing of outcome assessments

All visits are planned from the date of the first injection and are performed at week 7, 9, 13, 17, 21, and 27.

All irregularities are recorded as protocol deviations, and allowed visit windows are within ± 2 weeks.

**SEMALCO** study Statistical Analysis Plan

EU CT NUMBER: 2023-503371-25-00

03.06.25 Edition: 1.0

Statistical Principles

Confidence intervals and P-values

Statistical significance will be assessed using an alpha level of 0.05, with two-sided testing and a 95%

confidence interval. There will be no adjustment for multiplicity, and no additional adjustments for

covariates, except baseline values, will be performed.

Adherence and protocol deviations

Adherence to the intervention was defined by no more than three missed consecutive injections or six missed

injections in total during the 26-week period. The un-blinded project nurses kept an electronic individual

injection schedule per patient, tracking the extent of exposure to the assigned treatment. Adherence to the

intervention will be presented in a table showing the distribution of injection percentages and the number

of therapy sessions. Protocol deviations will be presented in a table divided into the categories: study

procedure, eligibility, and randomisation.

Analysis populations

All analyses will be performed using the intention-to-treat principle on subjects who received at least one

dose of the trial compound (Wegovy® or placebo).

**Trial Population** 

Screening data

Screening data will be presented in the CONSORT flowchart.

Eligibility

Individuals aged 18-70, BMI ≥30, diagnosed with AUD according to ICD 10 and DSM-5, with an AUDIT score

>15 and at least six heavy drinking days in the past 30 days.\* Furthermore, no severe psychiatric-,

neurological- or somatic disease, history of alcohol withdrawal seizures, diabetes, other substance use

disorder, or concomitant pharmacotherapy against alcohol use disorder. Please see the protocol paper for

the full list of in- and exclusion criteria.<sup>22</sup>

03.06.25

Edition: 1.0

SEMALCO study Statistical Analysis Plan

EU CT NUMBER: 2023-503371-25-00

The 30-day period will be the 30 consecutive days with the biggest alcohol intake (most heavy drinking days#

and the largest amount of total alcohol intake) out of the 40 days prior to the evaluation, measured by the

TLFB method

Recruitment

Recruitment began on the 13<sup>th</sup> of June, 2023 and ended on the 14<sup>th</sup> of February, 2025. The last patient's last

visit is in medio August, 2025. All participants were recruited from the capital region of Copenhagen and the

region of Zealand, Denmark.

Withdrawal/Follow up

All participants who have withdrawn from the intervention and have been included for at least 12 weeks

were encouraged to participate in the final follow-up at week 26, including brain scans at the time of

withdrawal. Due to safety concerns, all participants were contacted by telephone during week 31 to evaluate

any side effects. Drop-out data will be presented in a Kaplan-Meier survival curve as a function of the number

of injections received (the week they dropped out).

Baseline Patient characteristics

Baseline characteristics will be descriptively summarised in a table assessed by the intervention.

List of baseline characteristics to be summarised:

Sex, No. (%)

Age, mean (SD)

Age group (+/- 40 years)

Education (lower secondary school, upper secondary school, vocational education + short-cycle higher

education, medium cycle higher education + higher education), No. (%)

Marital status (Cohabitation + married), No. (%)

Job status (yes, no), No. (%)

Previous treatment with a GLP-1 receptor agonist (yes, no), No. (%)

Previous pharmacological treatment for AUD (disulfiram, acamprosate, naltrexone, nalmefene), No.

(%)

AUDIT score, mean (SD)

AUDIT-C score, mean (SD)

ICD-10 number of diagnostic items (4,5,6), No. (%)

03.06.25

Edition: 1.0

SEMALCO study Statistical Analysis Plan

EU CT NUMBER: 2023-503371-25-00

- DSM-5 group (mild (2-3), moderate (4-5), severe (>5)), No. (%)

Heavy drinking days\*, mean (SD)

- Heavy drinking days group/randomisation strata\* (6-11, 12-17, 18-23, 24-30), No. (%)

Days without alcohol consumption (0-days)\*, mean (SD)

Total alcohol consumption (grams)\*, mean (SD)

Plasma PEth, mean (SD)

- WHO risk level (low, medium, High, very high), No. (%)

Weight (kilogram), mean (SD)

- Body mass index (BMI), mean (SD)

Plasma HbA1c, mean (SD)

\*The 30-day period will be the 30 consecutive days with the biggest alcohol intake (most heavy drinking days **and** the largest amount of total alcohol intake) out of the 40 days prior to the evaluation, measured by the TLFB method.

## **Analysis**

### Primary endpoint

The primary endpoint is the change in alcohol consumption, defined as the change in the percentage of heavy drinking days during a period of 30 consecutive days\*, from baseline to end of follow-up after 26 weeks, adjusted for baseline (expressed in percentage points (pp)). A heavy drinking day is defined as more than 60/48 grams (men/women) of alcohol in one day, measured with the validated timeline followback (TLFB) method.<sup>25</sup>

\*The 30-day period will be the 30 consecutive days with the biggest alcohol intake (most heavy drinking days and the largest amount of total alcohol intake) out of the 40 days prior to the evaluation, measured by the TLFB method.

## Secondary endpoints

Changes from baseline to last assessment after 26 weeks of treatment with semaglutide vs placebo in:

1. Total alcohol consumption (gram ethanol/last 30 consecutive days\*)

2. Number of days without alcohol consumption (last 30 consecutive days\*)

3. Change in drinks per day (last 30 consecutive days\*)

4. Time to relapse, defined as the time to first alcohol intake

5. Time to first heavy drinking day

Edition: 1.0

- 6. WHO alcohol risk levels (last 30 consecutive days\*)
- 7. Alcohol craving (PACS score)
- 8. Alcohol Use Disorder Identification Test (AUDIT) score
- 9. Alcohol Use Disorder Identification Test (AUDIT-C) score
- 10. Blood Phosphatidylethanol (PEth)
- 11. Fibrosis-4 (FIB4) score
- 12. Blood gamma-glutamyl transferase (GGT)
- 13. Blood alanine transaminase (ALT)
- 14. Blood mean corpuscular volume (MCV)
- 15. Plasma amylase
- 16. Plasma semaglutide
- 17. Body weight (kg)
- 18. Blood pressure (mmHg)
- 19. Pulse (PR)
- 20. Waist circumference (cm)
- 21. BMI
- 22. Glycaemic control parameters (HbA1c)
- 23. Drug Use Disorders Identification Test (DUDIT) score
- 24. WHO quality of life BREF (WHOQOL-BREF) score
- 25. Fagerströms Test for Nicotine Dependence score

#### Descriptive statistics

The number of cognitive behavioural sessions during the follow-up period will be described by treatment group in order to assess if the individuals in the two treatment groups received equal amounts of therapy, and including any self-selected post-intervention treatment undertaken by the participants, if any. Also, the change in the percentage of heavy drinking days during a period of 30 consecutive days\*, from baseline to end of follow-up after 26 weeks will be plotted against (a) the maximum semaglutide dose during the 26 weeks of treatment, and (b) the weight loss at the end of follow-up.

### Analysis methods

All continuous outcomes, i.e., change in metabolic parameters, weight, body composition parameters, alcohol use, etc. will be analysed using baseline adjusted ANCOVA. The two time to event outcomes (time to first alcohol intake and time to first heavy drinking day) will be analysed using Cox regression.

03.06.25

Edition: 1.0

SEMALCO study Statistical Analysis Plan

EU CT NUMBER: 2023-503371-25-00

We will use residual plots and gq-plots in combination with Wally plots<sup>26</sup> to validate the normality assumption

of the residuals. If the distributional assumption about normality of the residuals does not hold then we will

first see if a log-transform of the outcome will result in a model fit that does not appear to violate the

assumptions of normality. If the log-transform still does not hold, our next step will be to consider if the lack

of fit is caused by inflation, e.g. due to too many observations being zero. Should that be the case we will

replace the standard ANOVA model with a zero-inflated gaussian model for the analyses. Should none of

these approaches work we will use quantile regression and model the median outcome instead.

Missing data/sensitivity analysis

Missing data will be imputed with the use of multiple imputations in the mice package<sup>27</sup> in R software<sup>28</sup>,

method = "pmm" (predictive mean matching), and 100 imputed datasets. The missing baseline and endpoint

data will be imputed based on a linear imputation model based on all available repeated measures data for

the outcome in question. As a sensitivity analysis, the complete case analysis will be performed. For the

outcomes of heavy drinking days, total alcohol intake, and days without alcohol consumption two further

sensitivity analyses regarding the missing data mechanism will be conducted: 1) assume that all non-

observed individuals at 26 weeks have reverted to their pre-study drinking habit, and 2) assume that all non-

observed individuals at 26 weeks have halved their drinking compared to the value at baseline.

Subgroup analysis

We will perform the following subgroup analysis for the primary outcome (change in alcohol consumption)

and for the outcomes of total alcohol consumption and number of days without alcohol consumption:

Baseline heavy days (6-11, 12-17, 18-23, 24-30)

DSM-5 group (mild (2-3), moderate (4-5), severe (>5))

Tertiary analyses

Tertiary analyses will be conducted and reported in subsequent secondary publications:

Proteomic fingerprint

Brain imaging:

Brain alcohol cue-response (Blood oxygenation level-dependent signal (BOLD)) in reward-processing

brain regions (ventral and dorsal striatum, putamen, nucleus accumbens, and caudate), including

the septal area assessed by fMRI brain scans

Brain GABA levels (cortical, caudate, and putamen) assessed by MRS brain scans

03.06.25

Edition: 1.0

**SEMALCO** study Statistical Analysis Plan

EU CT NUMBER: 2023-503371-25-00

Resting state functional connectivity

Diffusion tensor imaging (DTI)

Harms

Safety data has been collected in the 26 weeks of inclusion and up until 5 weeks after termination of the

study for all individuals. The safety outcomes were classified as adverse events (AE), adverse reactions (AR),

serious adverse events (SAE), serious adverse reactions (SAR), and suspected unexpected serious adverse

reactions (SUSAR). All collected safety data will be summarized in a table with number of cases.

Statistical software

Statistical analyses will be performed using R.

Edition: 1.0

EU CT NUMBER: 2023-503371-25-00

# References

- 1. Carvalho AF, Heilig M, Perez A, Probst C, Rehm J. Alcohol use disorders. Lancet 2019;394(10200):781–92.
- 2. WHO. Global status report on alcohol and health 2018. 2018.
- 3. Gottlieb Hansen AB, Hvidtfeldt UA, Grønbaek M, et al. The number of persons with alcohol problems in the Danish population. Scand J Public Health 2011;39:128–36.
- 4. Kohn R, Saxena S, Levav I, Saraceno B. The treatment gap in mental health care. Bull World Health Organ 2004;82(11):858–66.
- 5. Askgaard G, Leon DA, Deleuran T, Tolstrup JS. Hospital admissions and mortality in the 15 years after a first-time hospital contact with an alcohol problem: a prospective cohort study using the entire Danish population. Int J Epidemiol 2020;49(1):94–102.
- 6. Connor JP, Haber PS, Hall WD. Alcohol use disorders. Lancet 2016;387(10022):988–98.
- 7. Borges G, Bagge C, Cherpitel C, Conner K, Orozco R, Rossow I. A meta-analysis of acute alcohol use and the risk of suicide attempt Guilherme. Psychol Bull 2017;47(5):949–57.
- 8. Witkiewitz K, Litten RZ, Leggio L. Advances in the science and treatment of alcohol use disorder. Sci Adv 2019;5(eaax4043):1–11.
- 9. Nutt DJ, King LA, Phillips LD. Drug harms in the UK: A multicriteria decision analysis. Lancet 2010;376:1558–65.
- 10. Carroll KM, Kiluk BD. Cognitive Behavioral Interventions for Alcohol and Drug Use Disorders: Through the Stage Model and Back Again. Psychol Addict Behav 2017;31(8):847–61.
- 11. Magill M, Ray LA. Cognitive-behavioral treatment with adult alcohol and illicit drug users: A metaanalysis of randomized controlled trials. J Stud Alcohol Drugs 2009;70(4):516–27.
- 12. Morgenstern J, Longabaugh R. Cognitive-behavioral treatment for alcohol dependence: A review of evidence for its hypothesized mechanisms of action. Addiction 2000;95(10):1475–90.
- 13. Shen WW. Anticraving therapy for alcohol use disorder: A clinical review. Neuropsychopharmacol Reports 2018;38(3):105–16.
- 14. Lyon J. More Treatments on Deck for Alcohol Use Disorder. JAMA 2017;317(22):2267.
- 15. Davies M, Færch L, Jeppesen OK, et al. Semaglutide 2·4 mg once a week in adults with overweight or obesity, and type 2 diabetes (STEP 2): a randomised, double-blind, double-dummy, placebocontrolled, phase 3 trial. Lancet 2021;397(10278):971–84.
- 16. Gabery S, Salinas CG, Paulsen SJ, et al. Semaglutide lowers body weight in rodents via distributed neural pathways. JCI Insight 2020;5(6).

Edition: 1.0

EU CT NUMBER: 2023-503371-25-00

- 17. Kastin AJ, Akerstrom V, Pan W. Interactions of Glucagon-Like Peptide-1 (GLP-1) with the Blood-Brain Barrier. J Mol Neurosci 2002;18:7–14.
- 18. Salinas CBG, Lu TTH, Gabery S, et al. Integrated Brain Atlas for Unbiased Mapping of Nervous System Effects Following Liraglutide Treatment. Sci Rep 2018;8(1):1–12.
- 19. Secher A, Jelsing J, Baquero AF, et al. The arcuate nucleus mediates GLP-1 receptor agonist liraglutide-dependent weight loss. J Clin Invest 2014;124(10):4473–88.
- 20. Klausen MK, Knudsen GM, Vilsbøll T, Fink-Jensen A. Effects of GLP-1 Receptor Agonists in Alcohol Use Disorder. Basic Clin Pharmacol Toxicol 2025;136(3):1–15.
- 21. Leggio L, Hendershot CS, Farokhnia M, et al. GLP-1 receptor agonists are promising but unproven treatments for alcohol and substance use disorders. Nat Med 2023;
- 22. Klausen MK, Kuzey T, Pedersen JN, et al. Does semaglutide reduce alcohol intake in Danish patients with alcohol use disorder and comorbid obesity? Trial protocol of a randomised, double-blinded, placebo-controlled clinical trial (the SEMALCO trial). BMJ Open 2025;15(1):1–10.
- 23. Bogenschutz MP, Ross S, Bhatt S, et al. Percentage of Heavy Drinking Days Following Psilocybin-Assisted Psychotherapy vs Placebo in the Treatment of Adult Patients With Alcohol Use Disorder.

  JAMA Psychiatry 2022;10016.
- 24. Hallgren KA, Witkiewitz K. Missing Data in Alcohol Clinical Trials: A Comparison of Methods. Alcohol Clin Exp Res 2013;37(12):2152–60.
- 25. Sobell L., Sobell M. "Alcohol consumption measures," in Assessing Alcohol Problems: A Guide for Clinicians and Researchers. 1995.
- 26. Ekstrøm CT. Teaching "Instant Experience" with Graphical Model Validation Techniques. Teach Stat 2014;36(1):23–6.
- 27. van Buuren S, Groothuis-Oudshoorn K. "mice: Multivariate Imputation by Chained Equations in R." J Stat Softw 2011;45(3):1–67.
- 28. R Core Team (2020). R: A Language and Environment for Statistical Computing. R Foundation for Statistical Computing, Vienna, Austria.